CLINICAL TRIAL: NCT06898567
Title: EFFECT OF BLOOD PRESSURE MEASUREMENT IN DIFFERENT POSITIONS ON BLOOD PRESSURE VALUES AND ANXIETY LEVELS IN PREGNANT WOMEN WITH PREECLAMPSIA
Acronym: PREECLAMPSIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Şerife Kelle Dikbaş, Specialist Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: PREECLAMPSIA; 29.01.2024 2024/06 (Registry Identifier: Üsküdar University Non-Interventional Research Ethics Committee approval)
Record Dates: First submitted 2025-03-08; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia; Blood Pressure Check (Hypertension Screening)
Keywords: Preeclampsia; Blood pressure; Hypertension; Anxiety; Position
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were divided into three groups and their blood pressures were measured in the left lateral, right lateral and semi-fowler positions.
  Left Lateral Position: The pregnant patient was lying in the left lateral position on the bed, her head supported by a pillow of medium height. The left arm to be measured was positioned at heart level and supported by a pillow underneath. Blood pressure was measured using the arm extended at a 45° angle to the body in the left lateral position. Considering that taking measurements from the right arm above the heart level may decrease blood pressure values, both measurements were taken only from the left arm.
  Right Lateral Position: The pregnant woman was placed in the right lateral position on the bed. Her head was supported by a pillow of medium height. The right arm to be measured was held at heart level and extended at a 45° angle to the body. Considering that taking measurements from the left arm above the heart level may decrease blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right Lateral Position (Experimental): The pregnant woman was placed in the right lateral position on the patient bed. Her head was supported by a medium-height pillow. The right arm to be measured was held at heart level and extended at a 45° angle to the body. Considering that taking measurements from the left arm above heart level could lower blood pressure values, both measurements were made only from the right arm.
  Interventions: Other: Right Lateral Position
- Left Lateral Position (Experimental): The pregnant patient was lying in the left lateral position on her bed, her head supported by a pillow of medium height. The left arm to be measured was positioned at heart level and supported by a pillow underneath. Blood pressure was measured using the arm extended at a 45° angle to the body in the left lateral position. Considering that taking measurements from the right arm above heart level may lower blood pressure values, both measurements were taken from the left arm only.
  Interventions: Other: Left Lateral Position
- Semi Fowler Position (45° Fowler) (Experimental): The pregnant woman was laid on her back at a 45° angle on the patient bed. Her head was supported with a medium-height pillow. The arm to be measured was held at heart level and supported with a pillow underneath to provide the appropriate position.
  Interventions: Other: Semi Fowler Position (45° Fowler)

INTERVENTIONS:
Other: Right Lateral Position — Participants rested for 10 minutes in a fully seated position, leaning their backs on a chair, without crossing their legs and placing their feet parallel to the floor. During this time, the arm to be measured was kept at heart level.
  Arms: Right Lateral Position
Other: Left Lateral Position — Left Lateral Position
  Arms: Left Lateral Position
Other: Semi Fowler Position (45° Fowler) — Semi Fowler Position (45° Fowler)
  Arms: Semi Fowler Position (45° Fowler)

SUMMARY:
Aim: This study examined the effects of blood pressure measurement in different positions on diastolic and systolic blood pressure values and anxiety levels in pregnant women diagnosed with preeclampsia.

Method: The study was conducted between March and June 2024 as a pre-test post-test quasi-experimental study with 96 pregnant women diagnosed with preeclampsia in the perinatology department of a training and research hospital. Participants were divided into three groups and their blood pressures were measured in the left lateral, right lateral and semi-Fowler positions. Data were collected using an introductory information form and the State Anxiety Scale.

DETAILED DESCRIPTION:
Aim: This study examined the effects of blood pressure measurement in different positions on diastolic and systolic blood pressure values and anxiety levels in pregnant women diagnosed with preeclampsia.

Method: The study was conducted between March and June 2024 as a pre-test post-test quasi-experimental study with 96 pregnant women diagnosed with preeclampsia in the perinatology department of a training and research hospital. Participants were divided into three groups and their blood pressures were measured in the left lateral, right lateral and semi-Fowler positions. Data were collected using an introductory information form and the State Anxiety Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being primigravida (first pregnancy),

  * Being in the third trimester of pregnancy,
  * Being between the ages of 18-45,
  * Being diagnosed with preeclampsia,
  * Having an arm circumference of less than 36 cm,
  * Having a history of hospitalization of at least 24 hours (in order to minimize anxiety, uncertainty, lack of information and disorientation related to hospitalization).

Exclusion Criteria:

* • Presence of a physical disability that would make it difficult to perform the positions included in the study (e.g. loss of extremity),

  * Presence of decompensated disease (e.g. eclampsia, pulmonary edema),
  * Presence of a history of cardiological disease,
  * Diagnosis of obstructive sleep apnea,
  * Presence of additional risk factors other than preeclampsia (e.g. threat of premature birth, placental anomalies).

Ages: 18 Months to 45 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — pregnancies
Enrollment: 96 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
blood pressure measurement | 4 month
  The effect of blood pressure measurement in different positions on diastolic and systolic blood pressure values in pregnant women diagnosed with preeclampsia will be examined. Measurement will be made with a blood pressure device. Systolic pressure and diastolic pressure will be measured in mmhg.
anxiety levels | 4 month
  The effects of blood pressure measurement in different positions on anxiety levels in pregnant women diagnosed with preeclampsia will be measured. The anxiety level will be measured with the state anxiety scale. The score obtained from the scale varies between 20 and 80. A high score indicates a high level of anxiety, a low score indicates a low level of anxiety. The same applies when interpreting scores according to percentile rank. In other words, a low percentile rank (1, 5, 10) indicates low anxiety. The average score level determined in applications varies between 36 and 41.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women's and Children's Diseases Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stergiou GS, Palatini P, Parati G, O'Brien E, Januszewicz A, Lurbe E, Persu A, Mancia G, Kreutz R; European Society of Hypertension Council and the European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. 2021 European Society of Hypertension practice guidelines for office and out-of-office blood pressure measurement. J Hypertens. 2021 Jul 1;39(7):1293-1302. doi: 10.1097/HJH.0000000000002843. No abstract available. PMID 33710173
- [Result] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752